CLINICAL TRIAL: NCT05989776
Title: Assessment and Improvement of Regional Information and Coordination Tools to Promote Access to Fertility Preservation
Brief Title: Increasing Access to Fertility Preservation for Women with Breast Cancer
Acronym: EVAPREF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Paul Sabatier of Toulouse (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut Claudius Regaud (Other); Réseau Onco-Occitanie (Unknown); Réseau ONCOPL (Unknown)
Responsible Party: Principal Investigator, Marie-Anne Durand, Researcher, University Paul Sabatier of Toulouse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-057
Record Dates: First submitted 2023-06-26; First posted 2023-08-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Fertility preservation; Information; Practitioner training; Social inequalities in health; Participatory approach; Combined intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Oncologists

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized stepped-wedge trial multi-site evaluating access to fertility preservation counseling over a 30-month period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Usual care information to fertility preservation counseling
- Intervention: informational brochure for patients and brief training for oncologists (Active Comparator): The intervention is based on information provided to different target populations, using a variety of media, including brochures and videos.
  Interventions: Behavioral: Informational brochure for patients and brief training for oncologists

INTERVENTIONS:
Behavioral: Informational brochure for patients and brief training for oncologists — For this randomized, stepped wedge trial, the investigators planned a mixed intervention that targets both health professionals and patients. This intervention will be carried out in its entirety thanks to the working groups made up of health professionals and expert patients that took place before the randomized trial. The intervention for health professionals consists of awareness training. They will be trained (or made aware) at different times, defined by randomization. The intervention for patients consists of a pictorial information brochure and tabular patient decision aid given by trained health professionals.
  Arms: Intervention: informational brochure for patients and brief training for oncologists

SUMMARY:
The EVAPREF project aims to increase access to fertility preservation by developing an approach to improve and evaluate existing information and coordination tools developed by the Pays-de-la-Loire and Occitanie Regional Cancer networks. First, the investigators will use a qualitative, iterative, user-centered and participatory approach to improve the current tools and create training content for the physicians who will use these tools. Second, the investigators will conduct a randomized stepped wedge trial of women under 40 newly treated with chemotherapy for breast cancer. The investigators will evaluate the rate of fertility preservation consultation before and after implementation of the improved tools, over a 30-month period from mid-2023 to the end of 2025. Finally, in a third step, the investigators will study their approach (context-sensitive implementation analysis) and provide key elements for its transferability to other contexts and in particular to other Regional Cancer networks in France.

DETAILED DESCRIPTION:
Background:

With the increase in the number of long-term survivors, interest is shifting from cancer survival to life and quality of life after cancer. These include consequences of long-term side effects of treatment, such as gonadotoxicity. Fertility preservation is becoming increasingly important in cancer management. International recommendations agree on the need to inform patients prior to treatments about the risk of fertility impairment and refer them to specialized centers to discuss fertility preservation. However, the literature reveals suboptimal access to fertility preservation on an international scale, and particularly in France, making information for patients and oncologists a potential lever for action. The overall goal is to improve access to fertility preservation and related consultations for women with breast cancer through the development and evaluation of a combined intervention targeting the diffusion of information for these patients and brief training for oncologists.

Methods:

First, the investigators will use a qualitative, iterative, user-centered and participatory approach to improve existing information tools and create training content for oncologists (Aim 1). Second, the investigators will conduct a randomized stepped-wedge trial evaluating rate of fertility preservation consultation over a 30-month period (Aim 2). The investigators will include 750 women aged 18 to 40 newly treated with chemotherapy for breast cancer at one of 6 participating centers. The primary outcome will be rate of fertility preservation consultation before and after using the combined intervention (informational brochure for patients and brief training for oncologists) and will be analyzed using linear regression models.Third, the investigators will analyze their approach (context-sensitive implementation analysis) and provide key elements for transferability to other contexts in France (Aim 3).

Discussion:

After transitioning to the combined intervention, the investigators will expect to observe an increase in access to fertility preservation consultation. Particular attention will be paid to the effect of this intervention on socially disadvantaged women, who are known to be at greater risk of inappropriate treatment. In addition, the user-centric design principles and participatory approaches used to optimize the acceptability, usability and feasibility of the combined intervention will likely enhance its impact, diffusion and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 40 years of age treated for newly diagnosed breast cancer and receiving chemotherapy.
* People who are able to read the study information poster and the fertility preservation information brochure in French, either alone or with help from a caregiver or relative or an interpreter.
* People with intellectual disability will be included as long as they are able able to read the study information poster and the fertility preservation information brochure in French alone or with help from a caregiver or relative or an interpreter..

Exclusion Criteria:

* People whose mental health status precludes participation in the study, as determined by the clinical team.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recourse to fertility preservation consultation before and after using the combined intervention | up to 18 mont post enrollment
  This information will be collected by each regional screening coordination center of the two participating regions from the medical records of patients

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Anne Durand, PhD, Principal Investigator — Université Toulouse III Paul Sabatier
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - Institut Claudius Regaud (IUCT-O), Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Addamiano MC, Joannes C, Fonquerne L, Morel C, Lauzeille D, Belkadi L, Empereur F, Grosclaude P, Bauvin E, Delpierre C, Lamy S, Durand MA. Increasing access to fertility preservation for women with breast cancer: protocol for a stepped-wedge cluster randomized trial in France. BMC Public Health. 2024 Jan 19;24(1):231. doi: 10.1186/s12889-024-17719-3. PMID 38243214